CLINICAL TRIAL: NCT02349685
Title: The Efficacy of the Culture Based Tailored Therapy for Helicobacter Pylori Eradication Comparing With the Traditional 2nd Line Rescue Therapy in Korean
Brief Title: The Efficacy of the Tailored Therapy Based on Antimicrobial Susceptibility for 2nd Eradication of H. Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1412/280-119
Record Dates: First submitted 2015-01-25; First posted 2015-01-29 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-08

CONDITIONS: Helicobacter Infection
Keywords: Helicobacter pylori; Personalized therapy; antimicrobial susceptibility; rescue therapy; culture
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 14 day bismuth based quadruple therapy (PBMT) group (Experimental): Proton pump inhibitor (PPI) regular dose b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d
  Interventions: Drug: 14 day PBMT group
- 14 day Moxifloxacin containing triple therapy (MEA) group (Experimental): PPI regular dose b.i.d., moxifloxacin 400 mg q.d., and amoxicillin 1g b.i.d.
  Interventions: Drug: 14 day MEA group
- 14 day tailored therapy group (Active Comparator): based on H. pylori culture and antimicrobial sensitivity, select the 2nd rescue regimen between 14 days of bismuth-based quadruple therapy or 14 days moxifloxacin-containing triple therapy according to antibiotics susceptibility.
  Interventions: Procedure: H. pylori culture and antimicrobial susceptibility test

INTERVENTIONS:
Procedure: H. pylori culture and antimicrobial susceptibility test — Antral and body biopsy specimens were evaluated separately. Organisms were identified as H. pylori by Gram staining, colony morphology, and positive oxidase, catalase, and urease reactions. Minimum inhibitory concentrations (MICs) were determined by the agar dilution method. Amoxicillin (Sigma Chemical Co., St. Louis, Mo.), clarithromycin (Abbott Laboratories, Abbott Park, Ill.), metronidazole (Sigma), tetracycline (Sigma) and moxifloxacin (Sigma) for the H. pylori isolates were examined by use of the serial twofold agar dilution method and the reference of susceptibility testing was according to the recommendations of the Clinical and Laboratory Standards Institute [amoxicillin (AMC), MIC ≥ 0.5 μg / ml; clarithromycin (CLA), MIC > 1.0 μ g / ml; metronidazole (MET), MIC > 8 μ g / ml; tetracycline (TC), MIC > 4 μ g / ml; and moxifloxacin (MOX), MIC > 1 μ g / ml).
  Arms: 14 day tailored therapy group
Drug: 14 day PBMT group — Rescue therapy using 14 day PBMT regimen [Proton pump inhibitor (PPI) regular dose b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d]
  Arms: 14 day bismuth based quadruple therapy (PBMT) group
Drug: 14 day MEA group — Rescue therapy using 14 day MEA regimen (PPI regular dose b.i.d., moxifloxacin 400 mg q.d., and amoxicillin 1g b.i.d.)
  Arms: 14 day Moxifloxacin containing triple therapy (MEA) group

SUMMARY:
As increasing the antibiotics resistance, the effectiveness of traditional Helicobacter pylori (H. pylori) therapies has been declined coincidently. In this study, the investigators evaluated the efficacy of H. pylori eradication between a personalized therapy for H. pylori infection based on the results of antibiotics resistance by using H. pylori culture and minimal inhibitory concentration (MIC) and the traditional 2nd rescue regimens, and the investigators analyzed the prevalence of the antibiotic resistance after 1st eradication of H. pylori in the tailored therapy group.

DETAILED DESCRIPTION:
The patients who had shown the evidence of persistent H. pylori infection after the 1st eradication were enrolled for this study. After giving the informed consent about the method and efficacy (ITT and PP analysis) of the traditional 2nd rescue therapy and the tailored therapy for H. pylori infection based on culture and MIC, the patients were classified into the three regimen group under the patient's agreement and underwent 2nd eradication [14 days bismuth-based quadruple therapy (Proton pump inhibitor (PPI) regular dose b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d.), 14 days moxifloxacin-containing triple therapy (PPI regular dose b.i.d., moxifloxacin 400 mg q.d., and amoxicillin 1g b.i.d.), or tailored therapy based on H. pylori culture and MIC (select the 2nd rescue regimen between 14 days of bismuth-based quadruple therapy or 14 days moxifloxacin-containing triple therapy according to antibiotics susceptibility)].This study was analyzed the success of eradication for enrolled participants retrospectively, however the patients were enrolled prospectively based on previous study about antimicrobial susceptibility test for H. pylori in Korea.

ELIGIBILITY:
Inclusion Criteria:

* The patients who proved a failure of 1st eradication of H. pylori with Proton pump inhibitor based triple therapy (PPI bid + amoxacillin 1g b.i.d + Clarithromycin 500 mg b.i.d) or sequential therapy (initial 5-day therapy with a combination of PPI b.i.d and amoxicillin 1g b.i.d, followed by 5 days of PPI b.i.d., clarithromycin 500mg b.i.d., and metronidazole 500mg t.i.d) following three methods

  1. positive rapid urease test (CLOtest)
  2. histologic evidence of H. pylori by modified Giemsa staining
  3. positive 13C-Urea breath test
* Male and female Korean Adult (Aged ≥ 18 years)

Exclusion Criteria:

* Patients who received two or more eradication therapy for H. pylori infection
* H. pylori eradication failure because of poor compliance
* the administration of antibiotics or the consumption of bismuth salts within 4 weeks or the administration of a proton pump inhibitor (PPI) within 2 weeks
* Advanced gastric cancer or other malignancy
* Abnormal liver function or liver cirrhosis
* Abnormal renal function or chronic kidney disease
* Other severe concurrent diseases
* Previous allergic reactions to the study drugs
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph. D, Principal Investigator — Seoul National University Bundang Hospital

REFERENCES:
- [Derived] Kwon YH, Kim N, Lee JY, Choi YJ, Yoon K, Nam RH, Suh JH, Lee JW, Lee DH. Comparison of the efficacy of culture-based tailored therapy for Helicobacter pylori eradication with that of the traditional second-line rescue therapy in Korean patients: a prospective single tertiary center study. Scand J Gastroenterol. 2016 Mar;51(3):270-6. doi: 10.3109/00365521.2015.1095352. Epub 2015 Oct 9. PMID 26452405

RESULTS

PARTICIPANT FLOW:
Groups:
- 14 Day PBMT Group: Proton pump inhibitor (PPI) regular dose b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d
  14 day PBMT group: Rescue therapy using 14 day PBMT regimen [Proton pump inhibitor (PPI) regular dose b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d]
- 14 Day MEA Group: PPI regular dose b.i.d., moxifloxacin 400 mg q.d., and amoxicillin 1g b.i.d.
  14 day MEA group: Rescue therapy using 14 day MEA regimen (PPI regular dose b.i.d., moxifloxacin 400 mg q.d., and amoxicillin 1g b.i.d.)
- 14 Day Tailored Therapy Group: based on H. pylori culture and MIC, select the 2nd rescue regimen between 14 days of bismuth-based quadruple therapy or 14 days moxifloxacin-containing triple therapy according to antibiotics susceptibility.
Period: Overall Study
Arm/Group | 14 Day PBMT Group | 14 Day MEA Group | 14 Day Tailored Therapy Group
Started | 89 | 89 | 41
Completed | 84 | 87 | 37
Not Completed | 5 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 14 Day PBMT Group | 14 Day MEA Group | 14 Day Tailored Therapy Group | Total
Number analyzed (Participants) | 89 | 89 | 41 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 52 | 27 | 128
  >=65 years | 40 | 37 | 14 | 91
Age, Continuous [Mean (Full Range); unit: years] | 55.7 [18 to 74] | 59.2 [25 to 75] | 54.5 [29 to 75] | 54.5 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 53 | 25 | 121
  Male | 46 | 36 | 16 | 98
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 89 | 89 | 41 | 219

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Arm/Group With Successful H. Pylori Eradication
Description: the efficacy of H. pylori eradication between a personalized therapy for H. pylori infection based on the results of antibiotics resistance by using H. pylori culture and minimal inhibitory concentration (MIC) and the traditional 2nd rescue regimens.
  The eradication rate was evaluated by intention to treat (ITT)
Time Frame: 6 weeks after completion of eradication
Measure: Number; unit: participants
Groups:
- 14 Day Tailored Therapy Group: based on H. pylori culture and MIC, select the 2nd rescue regimen between 14 days of bismuth-based quadruple therapy or 14 days moxifloxacin-containing triple therapy according to antibiotics susceptibility.
  H. pylori culture and antimicrobial susceptibility test: Antral and body biopsy specimens were evaluated separately. Organisms were identified as H. pylori by Gram staining, colony morphology, and positive oxidase, catalase, and urease reactions. Minimum inhibitory concentrations (MICs) were determined by the agar dilution method. Amoxicillin (Sigma Chemical Co., St. Louis, Mo.), clarithromycin (Abbott Laboratories, Abbott Park, Ill.), metronidazole (Sigma), tetracycline (Sigma) and moxifloxacin (Sigma) for the H. pylori isolates were examined by use of the serial twofold agar dilution method and the reference of susceptibility testing was according to the recommendations of the Clinical and Laboratory Standards Institute.
Arm/Group | 14 Day PBMT Group | 14 Day MEA Group | 14 Day Tailored Therapy Group
Number analyzed (Participants) | 89 | 89 | 41
participants | 67 | 63 | 36

2. Secondary Outcome: Number of Participants in Each Arm/Group With Successful H. Pylori Eradication
Description: the efficacy of H. pylori eradication between a personalized therapy for H. pylori infection based on the results of antibiotics resistance by using H. pylori culture and minimal inhibitory concentration (MIC) and the traditional 2nd rescue regimens.
  The eradication rate was evaluated by per-protocol analysis (PP)
Time Frame: 6 weeks after completion of eradication
Measure: Number; unit: participants
Arm/Group | 14 Day PBMT Group | 14 Day MEA Group | 14 Day Tailored Therapy Group
Number analyzed (Participants) | 84 | 87 | 37
participants | 67 | 63 | 37

ADVERSE EVENTS:
Arm/Group | 14 Day PBMT Group | 14 Day MEA Group | 14 Day Tailored Therapy Group
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/87 | 0/37
Other Adverse Events (participants affected / at risk) | 0/84 | 0/87 | 0/37

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other